CLINICAL TRIAL: NCT04246060
Title: Multicentre, Ambispective, Observational, Real Life Study to Assess the Quality of Life Effectiveness of Extended Release (ER) Oral Cysteamine Therapy (Procysbi) in Belgian Patients Suffering From Nephropathic Cystinosis
Brief Title: Observational Study to Assess the Quality of Life in Nephropathic Cystinosis Patients
Acronym: PROREAL
Status: Enrolling by invitation | Type: Observational
Sponsor: Chiesi SA/NV (Other)
Responsible Party: Sponsor
Other Study IDs: CHIESI-NIS-003
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Nephropathic Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — Cysteamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Patients on extended release cysteamine treatment at study enrollment
  Interventions: Drug: Cysteamine Bitartrate
- Cohort 2: Patients switching from immediate release cysteamine to extended release cysteamine during the study
  Interventions: Drug: Cysteamine Bitartrate
- Cohort 3: Patients remaining on immediate release cysteamine treatment
  Interventions: Drug: Cysteamine Bitartrate

INTERVENTIONS:
Drug: Cysteamine Bitartrate — ERT

SUMMARY:
Most of the real world evidence data related to efficacy of cysteamine therapy is retrospective. This study is a ambispective study to investigate the impact of cystine depletion therapy on the quality of life of patients and their parents.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of nephropathic cystinosis
* Undergoing cystine depletion therapy with oral cysteamine
* Signature of informed concent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Belgian nephropathic cystinosis patients.
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
to descriptively assess the change from baseline and percent change from baseline in the quality of life overall summary sores at 12 months in switch cohort | 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (7):
  - UZA, Antwerp
  - HUDERF, Brussels
  - UCL Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHC, Liège
  - CHU, Liège